CLINICAL TRIAL: NCT01596738
Title: Tranexamic Acid in Patients Receiving Primary and Isolated On-pump CABG With Premature Clopidogrel Cessation to Reduce Postoperative Bleeding and Transfusion
Brief Title: Tranexamic Acid in On-pump CABG With Premature Clopidogrel Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Li Lihuan (Other)
Responsible Party: Sponsor-Investigator, Li Lihuan, Professor and director of the department of anesthesiology and critical care, NCCD, PUMC & CAMS, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fuwai2008
Record Dates: First submitted 2012-05-05; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Graft
Keywords: Coronary Artery Disease; Coronary Artery Bypass Graft; Platelet Aggregation Inhibitors; Tranexamic Acid
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid group (Experimental): 1. Tranexamic acid 50mg/ml, 15 mg/kg intravenous after anesthetic induction
  2. Tranexamic acid 50mg/ml, 15 mg/kg intravenous after neutralization
  Interventions: Drug: Tranexamic Acid
- Placebo group (Placebo Comparator): 1. Equivalent volume of saline, equal to that of 50mg/ml tranexamic acid at the dosage of 15mg/kg, intravenous after anesthetic induction
  2. Equivalent volume of saline, equal to that of 50mg/ml tranexamic acid at the dosage of 15mg/kg, intravenous after neutralization
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic Acid — 1. Tranexamic acid 50mg/ml, 15 mg/kg intravenous after anesthetic induction
  2. Tranexamic acid 50mg/ml, 15 mg/kg intravenous after neutralization
  Arms: Tranexamic Acid group
Drug: Saline — 1. Equivalent volume of saline, equal to that of 50mg/ml tranexamic acid at the dosage of 15mg/kg, intravenous after anesthetic induction
  2. Equivalent volume of saline, equal to that of 50mg/ml tranexamic acid at the dosage of 15mg/kg, intravenous after neutralization
  Arms: Placebo group

SUMMARY:
The use of platelet aggregation inhibitors, including aspirin and clopidogrel, has become a standard management strategy for patients with acute coronary syndrome. On this background, an increasing percentage of patients presenting for surgical coronary revascularization is the subject to irreversible platelet inhibition.

Tranexamic acid is a widely used antifibrinolytic agent, and is a promising substitute for aprotinin when the latter has been suspended in 2007.The release of plasmin during CPB activates fibrinolysis and may contribute to platelet dysfunction. Pharmacological inhibition of the fibrinolytic system may therefore ameliorate platelet dysfunction and fibrinolysis after CPB and decrease postoperative bleeding. Tranexamic acid prevents plasmin formation and inhibits fibrinolysis.

Many studies and meta-analyses have shown a reduction in postoperative bleeding and transfusion requirements of this antifibrinolytic drug in cardium revascularization surgery. Unfortunately the preoperative antiplatelet therapy was either neglected or obscure. Few studies specify the time between the last clopidogrel ingestion and surgery.Several studies were keen on the blood loss and allogeneic transfusion in patients who received their last clopidogrel or asprin within 7 days prior to coronary artery bypass grafting. Concerning the secession of aprotinin and the increasing proportion of patients with persistence on clopidogrel until their surgery, evolutional work is expected, especially in the eastern population.

The purpose of this study is to assess the effect of tranexamic acid in patients with clopidogrel and asprin ingestion less than 7 days prior to surgery. The working hypothesis is that tranexamic acid would reduce bleeding and transfusion requirements in this specific population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-85 years undergoing primary and isolated on-pump CABG
* Last ingestion of clopidogrel and aspirin within 7 days preoperatively

Exclusion Criteria:

* Previous cardiac surgery
* Hematocrit <33%
* Platelet count <100,000/ml
* Allergy to tranexamic acid
* Recruited in other studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Allogeneic erythrocyte, volume transfused | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Total volume of allogeneic erythrocyte transfused, from the beginning of the operation until discharge
Allogeneic erythrocyte, percentage exposed | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The percentage of patients exposed to allogeneic erythrocyte, from the beginning of the operation until discharge

SECONDARY OUTCOMES:
Blood loss | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The total volume of chest drainage from the end of the operation until the removal of the drainage tube
Major bleeding | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The incidence of major bleeding according to the CURE definition
Reoperation | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The incidence of reoperation for excessive bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Lihuan Li, M.D., Principal Investigator — Cardiovascular Institute and Fuwai Hospital, NCCD, PUMC & CAMS
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, Beijing, China